CLINICAL TRIAL: NCT06078384
Title: Adjuvant Pembrolizumab and Chemotherapy or Surveillance in Early Triple Negative breAst Cancer With High Stromal Tumor-infiltrating Lymphocytes (TILs) Score
Brief Title: Pembrolizumab and Chemotherapy Treatment or no Treatment Guided by the Level of TILs in Resected Early-stage TNBC
Acronym: ETNA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: MSD France (Industry); SOLTI Breast Cancer Research Group (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); Vall Hebron Insitut Recerca (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-BCG-2213; 2023-504620-26-00 (Other: EU Clinical Trials Register)
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Triple-negative Breast Cancer
Keywords: Breast cancer; De-escalation; Immunotherapy; Chemotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — pembrolizumab; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Cohort of patients with T1b/c N0 M0 TNBC aged > 40 years with 30% ≤ sTILs < 50% and those aged ≤ 40 years with 30% ≤ sTILs < 75%: Pembrolizumab will be administered at a fixed dose of 200 mg every 3 weeks (Q3W), with a total of 9 cycles and Paclitaxel 80 mg/m² weekly for 12 cycles at adjuvant phase of the treatment; Cohort of patients with T1b/c N0 M0 TNBC aged > 40 years and sTILs ≥ 50% and those aged ≤ 40 years with sTILs ≥ 75%: No treatment will be administered. These patients will undergo standard surveillance every 6 months according to local practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1-Pembrolizumab plus Paclitaxel (Experimental): Pembrolizumab will be administered at a fixed dose of 200 mg every 3 weeks (Q3W), with a total of 9 cycles and Paclitaxel 80 mg/m² weekly for 12 cycles
  Interventions: Drug: Pembrolizumab 25 mg/ml; Drug: Paclitaxel injection
- Cohort 2-Observation (No Intervention): No treatment will be administered, patients will undergo standard surveillance every 6 months according to local practice.

INTERVENTIONS:
Drug: Pembrolizumab 25 mg/ml — Pembrolizumab drug product is a sterile-filtered liquid and is aseptically filled into single-use vials.
  The vials contain 4 mL of sterile solution for IV infusion.
  Other Names: keytruda
  Arms: Cohort 1-Pembrolizumab plus Paclitaxel
Drug: Paclitaxel injection — Injectable solution for IV administration. Dose of 80 mg/m² weekly.
  Other Names: Taxol
  Arms: Cohort 1-Pembrolizumab plus Paclitaxel

SUMMARY:
Triple-negative breast cancer (TNBC) is a group of tumors that occurs mainly in young, premenopausal women and accounts for 10-20% of breast cancers. Over the past decade, the incidence of women diagnosed with early-stage TNBC has significantly increased due to the widespread use of screening mammography. Treatment of patients with localized TNBC mainly involves surgery and (neo)adjuvant chemotherapy with or without radiotherapy. However, the benefit of chemotherapy may be controversial in patients with early-stage TNBC defined by small size and absence of lymph node involvement, and with significant tumor lymphocyte infiltration.

The ETNA study is a phase II trial designed to evaluate a chemotherapy de-escalation strategy in patients with TNBC T1b/c N0M0 and stromal TILs (sTILs) ≥ 30%. ETNA comprises two cohorts defined according to the level of TILs and the age of patients. Patients aged > 40 years with 30% ≤ sTILs < 50% and those aged ≤ 40 years with 30% ≤ sTILs < 75% will be included in the cohort 1 and will receive adjuvant pembrolizumab 200 mg every three weeks for 9 cycles and Paclitaxel 80 mg/m² weekly for 12 cycles. Patients aged > 40 years with sTILs ≥ 50% and those aged ≤ 40 years with sTILs ≥ 75% will be included in cohort 2 and will not receive adjuvant treatment, they will undergo standard surveillance every six months.

DETAILED DESCRIPTION:
(Neo)adjuvant chemotherapy in breast cancer is associated to long-term persistent QoL deterioration in patients with early breast cancer, with a greater negative impact in patients that were premenopausal at diagnosis. Because triple negative breast cancer (TNBC), which accounts for 10-20% of breast cancers, presents a poorer prognosis as compared to the other subtypes, international guidelines endorse the use of adjuvant chemotherapy from TNBC tumors measuring > 5 mm. Nevertheless, a number of retrospective studies have reported excellent prognosis for patients with small, lymph node-negative and high TILs TNBC, even without chemotherapy, with 5-year overall survival (OS) of 98%. Findings from multiple data sets consistently demonstrated that TILs represent a robust prognostic and predictive biomarker in early-stage TNBC, being now the first biological prognostic marker for TNBC included in several international guidelines for early-stage disease, such as 2019 St Gallen consensus conference and European Society for Medical Oncology (ESMO) Guidelines for early-stage breast cancer.

In clinical practice, oncologists have taken different approaches in patients with stage I TNBC. While some have de-escalated anthracyclines, other did not held back on the standard chemotherapy options with anthracyclines, taxanes, and cyclophosphamide. Based on unpublished data from the TNBC pooled analysis with sTILs on 2211 patients not treated by systematic therapy, performed at Gustave Roussy, the 5-year distant disease free-survival (DDFS) is 87%, 91%, and 93% for those with stage I and sTILs ≥ 30%, 50%, and 75%, respectively. Given these compelling findings from historical observations, it is reasonable to anticipate that the absolute benefit of chemotherapy would be modest among these patients as their tumors generally exhibit a favorable prognosis, resulting in reduced benefits with the use of adjuvant chemotherapy.

ETNA is a phase II, multicenter, biomarker-driven study that is designed to characterize the clinical course of patients with stage I TNBC and sTILs ≥ 30%.

ETNA includes patients with stage I and sTILs ≥ 30% TNBC in 2 cohorts:

* Cohort 1 will include patients age > 40 years with 30% ≤ sTILs < 50% and those aged ≤ 40 years with 30% ≤ sTILs < 75%. Patients will receive 9 cycles of adjuvant pembrolizumab 200 mg every three weeks for 9 cycles and Paclitaxel 80 mg/m² weekly for 12 cycles.
* Cohort 2 will include patients aged > 40 years with sTILs ≥ 50% and those aged ≤ 40 years with sTILs ≥ 75% who will undergo standard surveillance (no adjuvant systemic treatments).

ELIGIBILITY:
Inclusion Criteria:

1. Understand, sign, and date the written informed consent form prior to any protocol- specific procedures performed,
2. Men and women aged ≥ 18 years,
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1,
4. Histologically confirmed and radically removed pT1b/c N0M0 TNBC as defined according to AJCC TNM stage-8th version,

   * Histologically documented TNBC (negative HER2, ER, and PgR status). HER2 negativity is defined by local laboratory assessment using in situ hybridization and immunohistochemistry assays as per ASCO/CAP criteria and ER/PgR negativity is defined by local laboratory assessment < 10% using immunohistochemistry assays,
   * Bilateral and/or multifocal primary tumor is allowed and the tumor with the most advanced T stage should be used to asses for eligibility. If multifocal tumor, a pathologic confirmation of TNBC is required for each focus,
5. Adequately excised breast cancer: subjects must have undergone either breast- conserving surgery or mastectomy/nipple- or skin-sparing mastectomy.

   * For subjects who undergo breast-conserving surgery, the margins of the resected specimen must be histologically free of invasive tumor and ductal carcinoma in situ (DCIS) as determined by the local pathologist. Reresections to ensure no ink on tumor margins are allowed. Subjects with margins positive for lobular carcinoma in situ (LCIS) are eligible without additional resection.
   * For subjects who undergo mastectomy/nipple- or skin-sparing mastectomy, margins must be free of gross residual tumor. It is recommended that subjects should have a negative microscopic margin in accordance with local pathology protocol,
6. Have had sentinel lymph node biopsy (SLNB) and/or axillary lymph node dissection (ALND) for evaluation of pathologic nodal status.

   Axillary nodal dissection(s) should yield a total of at least six nodes (including the axillary lymph nodes resected at the SLNB plus the lymph nodes collected at the axillary nodal dissection),
7. At least 4 weeks but no more than 12 weeks between definitive breast surgery (or the last surgery with curative intent if additional resection is required for breast cancer) and treatment initiation for cohort 1 and no more than 12 weeks for cohort 2,
8. Centrally assessed TILs score from surgical formalin-fixed paraffin embedded (FFPE) tumor sample, using an H&E stained diagnostic digital slide, according to the most recent International TILs Working Group guidelines,

   * Cohort 1 will include patients aged > 40 years with 30% ≤ sTILs < 50% and those aged

     * 40 years with 30% ≤ sTILs < 75%
   * Cohort 2 will include patients aged > 40 years with sTILs ≥ 50% and those aged ≤ 40 years with sTILs ≥ 75%
9. Women of childbearing potential have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication for cohort 1 and within 7 days of inclusion for cohort 2,
10. Women of childbearing potential must agree to use protocol-specified method(s) of contraception for 3 years after patient inclusion. Men subjects who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception during trial treatments and for at least 6 months after the last dose of trial treatments.

    Females of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year,
11. Patients affiliated to the social security system (or equivalent)- France only,
12. Patient is willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up.

    Additional inclusion criteria for subjects of cohort 1:
13. Left ventricular ejection fraction (LVEF) of ≥ 50% as assessed by echocardiogram or cardiac scintigraphy,
14. Demonstrate adequate organ function within 7 days of inclusion

    * Absolute Neutrophil Count (ANC) ≥ 1,500 /µL
    * Platelets ≥ 100,000 /µL
    * Hemoglobin ≥ 9 g/dL
    * Creatinine clearance ≥ 30 mL/min for subject with creatinine levels > 1.5 x institutional upper limit of normal (ULN)
    * Total bilirubin ≤ 1.5 x ULN or direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
    * Albumin ≥ 3.0 g/dL
    * Lactate dehydrogenase (LDH) < 2.5 X ULN
    * International normalized ratio/partial thromboplastin time (INR/PTT) ≤ 1.5 x ULN (unless subject is receiving anticoagulant therapy as long as prothrombin time (PT) or PTT is within therapeutic range of intended use of anticoagulants)
    * Thyroid stimulating hormone (TSH), free T4 (FT4), and free T3 (FT3) within normal ranges
    * Cortisol at 8 AM within normal ranges
    * Lipase and amylase < 3 ULN
    * Fasting plasma glucose ≤ 120 mg/dl or 6.7 mmol/L
    * Troponin within normal range

Exclusion Criteria:

1. History of invasive malignancy ≤ 3 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer,
2. Having received prior chemotherapy or targeted therapy within the past 12 months,
3. Has a prior history of DCIS and/or LCIS that was treated with any form of systemic, hormonal therapy, or radiotherapy to the ipsilateral breast; subjects who had their DCIS/LCIS treated only with surgery and/or contralateral DCIS treated with radiotherapy are allowed to enter the study,
4. Having received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agents or with an agent directed to another co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137),
5. Treatment with systemic immunostimulatory agents (including, but not limited to, interferons, interleukin-2) within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to inclusion,
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive medications (including prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] alpha agents) within 7 days prior to inclusion:

   * Subjects who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study
   * The use of inhaled corticosteroids and mineralocorticoids is allowed,
7. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment; subjects with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are eligible if:

   * Rash must covers <10% of body surface area.
   * Disease is well controlled at baseline and requires only low-potency topical Corticosteroids and no acute exacerbations requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or oral corticosteroids occurred within the previous 12 months,
8. Has a known history of Human Immunodeficiency Virus (HIV),
9. Prior allogeneic stem cell or solid organ transplant,
10. Has a known history of active Bacillus Tuberculosis,
11. Patients with any other disease or illness which requires hospitalisation or is incompatible with the trial treatment are not eligible,
12. Pregnant women or breastfeeding or expecting to conceive within the projected duration of the study, from the inclusion visit until the end of the 3 years follow up. Men subjects who engage in heterosexual intercourse and refuse to use protocol-specified method(s) of contraception during trial treatments and for at least 6 months after the last dose of trial treatments,
13. Patients unable to comply with trial obligations for geographic, social, or physical reasons, or who are unable to understand the purpose and procedures of the trial,
14. Person deprived of their liberty or under protective custody or guardianship,
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

    Additional non-inclusion criteria for subjects of cohort 1:
16. Has cardiac dysfunction as defined by any of the following prior to inclusion:

    * History of NCI-CTCAE v5.0 Grade > 3 symptomatic congestive heart failure or New York Heart Association (NYHA) criteria Class II,
    * Angina pectoris requiring anti-anginal medication, serious cardiac arrhythmia not controlled by adequate medication, severe conduction abnormality, or clinically significant valvular disease,
    * Significant symptoms (≥ Grade 2) relating to left ventricular dysfunction or cardiac ischemia,
17. Has a known hypersensitivity (≥ Grade 3) to the components of the study therapy or its analogs,
18. Has received a live vaccine or live-attenuated vaccine within 30 days of the first dose of study treatment,
19. Concurrent active Hepatitis B virus (HBV; defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (HCV; defined as anti-HCV Ab positive and detectable HCV RNA) infection,
20. Severe infections within 4 weeks prior to initiation of study treatment, including, hospitalization for complications of infection, bacteremia, or severe pneumonia,
21. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment; subjects receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection) are eligible,
22. Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment or anticipation of need for a major surgical procedure during study treatment,
23. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has a current pneumonitis/interstitial lung disease,
24. Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 4 weeks of the first dose of treatment in this current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Distant disease-free survival (DDFS) | 5 year
  Distant disease-free survival is defined as the delay between date of inclusion and distant tumor relapse, second cancer, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Invasive disease-free survival (IDFS) | From inclusion up to 5 year
  Invasive disease-free survival is defined as the delay between date of inclusion and invasive breast tumor recurrence, distant recurrence, second cancer, or death from any cause, whichever occurs first.
Distant recurrence-free survival (DRFS) | From inclusion up to 5 year
  Distant recurrence-free survival is defined as the delay between date of inclusion and distant recurrence of breast cancer or death from any cause, whichever occurs first.
Overall survival (OS) | From inclusion to death from any cause, up to 5 year
  The overall survival is the length of time from inclusion that patients enrolled in the study are still alive.
Incidence of Adverse Events | Throughout study completion, up to 5 year
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, every 3 weeks for 6 months then every 6 months up to 5 years
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Breast cancer module (QLQ-BR23) | At baseline, every 3 weeks for 6 months then every 6 months up to 5 years
  This EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR23 contains 23 items incorporating five multi-item scales to assess systemic therapy side effects, arm symptoms, breast symptoms, body image and sexual functioning. In addition, single items assess sexual enjoyment, hair loss and future perspective. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. For all items but sexual functioning and sexual enjoyment, higher scores indicate more severe symptoms.
Quality of Life Questionnaire - Cancer-related fatigue (QLQ-FA12) | At baseline, every 3 weeks for 6 months then every 6 months up to 5 years
  This EORTC cancer related fatigue questionnaire is intended to supplement the QLQ-C30.
  The QLQ-FA12 contains 12 items organized in three subscales: physical fatigue (5 items), emotional fatigue (3 items), and cognitive fatigue (2 items). The remaining two items serve as global indicators for interference of fatigue with daily activities and social sequelae of fatigue. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale with higher scores indicating greater degree of fatigue.
Hospital anxiety and depression scale (HADS) | At baseline, every 3 weeks for 6 months then every 6 months up to 5 years
  The HADS is a 14 items questionnaire: 7 items related to anxiety and 7 items related to depression scored on a scale. Scores for items in each subscale of the HADS are summed to produce an anxiety score (HADS-A) or a depression score (HADS-D), or can be added to produce a total score corresponding to emotional distress (HADS-T). Each item is rated on a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), for a total score ranging from 0-21 for each subscale. The entire scale (emotional distress) range from 0 to 42, with higher scores indicating more distress.

CONTACTS AND LOCATIONS:
Overall Officials: Elie Rassy, MD, Principal Investigator — Gustave Roussy, Villejuif, France; Barbara Pistilli, MD, Principal Investigator — Gustave Roussy, Villejuif, France; Mafalda Oliveira, MD, Principal Investigator — HOSPITAL VALL D'HEBRÓN, Barcelona, Spain
Locations (44):
- France (30):
  - CHU Amiens Picardie_Site Sud, Amiens
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre François Baclesse, Caen
  - Pôle Santé Republique, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges-François Leclerc, Dijon
  - Hôpital Franco-Britannique-Fondation Cognacq-Jay, Levallois-Perret
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Hopital Privé Jean Mermoz, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut régional du Cancer de Montpellier, Montpellier
  - Hôpital privé du confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU de Nîmes, Nîmes
  - Centre Hospitalier de Pau, Pau
  - Hôpital Privé des côtes d'Armor, Plérin
  - Hôpital NOVO, Pontoise
  - Centre Hospitalier de Cornouaille, Quimper
  - Clinique La Croix du Sud, Quint-Fonsegrives
  - Institut Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - CHU de Saint Etienne, Saint-Etienne
  - Institut Claudius Regaud, Toulouse
  - CHU Bretonneau, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Spain (14):
  - Hospital General Universitario Dr.Balmis, Alicante
  - Ico Badalona, Badalona
  - Hospital Vall D'Hebrón, Barcelona
  - Hospital Clinico Universitario Virgen de La Arrixaca, El Palmar
  - Hospital Universitario Clinico San Cecilio, Granada
  - Ico Hospitalet, L'Hospitalet de Llobregat
  - Complejo Asistencial Universitario de Leon, León
  - Hu Arnau de Vilanova Lleida, Lleida
  - Hospital Ramon Y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Sant Joan de Reus, Reus
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clínico Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.